CLINICAL TRIAL: NCT00092040
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Multicenter Study to Evaluate and Compare the Effects of Alendronate and Risedronate on Bone Mineral Density in Postmenopausal Women With Osteoporosis; A 12 Month Extension to: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Multicenter Study to Evaluate and Compare the Effects of Alendronate and Risedronate on Bone Mineral Density in Postmenopausal Women With Osteoporosis
Brief Title: A Study and 12 Month Extension to Evaluate Two Investigational Drugs in Postmenopausal Women With Osteoporosis (MK-0217-907)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-907; 2004_019
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217, alendronate sodium/Duration of Intervention: 12 mo
Drug: Comparator: risedronate / Duration of Intervention: 12 mo

SUMMARY:
The purpose of this study and 12 month extension is to evaluate the effects of two investigational drugs on osteoporosis in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with osteoporosis

Exclusion Criteria:

* Any known allergy to the study drug

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 2003-03-18 (Actual); Primary Completion 2004-10-18 (Actual); Study Completion 2005-09-28 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline in hip trochanter bone mineral density (BMD)

SECONDARY OUTCOMES:
Mean percent change from baseline in PA lumbar spine, total hip, and femoral neck BMD

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Reid DM, Hosking D, Kendler D, Brandi ML, Wark JD, Weryha G, Marques-Neto JF, Gaines KA, Verbruggen N, Melton ME. Alendronic acid produces greater effects than risedronic acid on bone density and turnover in postmenopausal women with osteoporosis : results of FACTS -international. Clin Drug Investig. 2006;26(2):63-74. doi: 10.2165/00044011-200626020-00002. PMID 17163237
- [Background] Reid DM, Hosking D, Kendler D, Brandi ML, Wark JD, Marques-Neto JF, Weryha G, Verbruggen N, Hustad CM, Mahlis EM, Melton ME. A comparison of the effect of alendronate and risedronate on bone mineral density in postmenopausal women with osteoporosis: 24-month results from FACTS-International. Int J Clin Pract. 2008 Apr;62(4):575-84. doi: 10.1111/j.1742-1241.2008.01704.x. PMID 18324951